CLINICAL TRIAL: NCT04792151
Title: PHP TIES: Pilot Transdiagnostic Treatment Implementation and Effectiveness Study for Youth Emotional Disorders in a Partial Hospitalization Program
Brief Title: Youth PHP Pilot Transdiagnostic Treatment Implementation and Effectiveness Study
Acronym: PHP TIES
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Psychological Foundation (Other); Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Other Study IDs: 20-2566
Record Dates: First submitted 2021-01-15; First posted 2021-03-10 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Emotional Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PHP Youth: Youth ages 6-17 receiving standard of care treatment (i.e., transdiagnostic intervention for emotional disorders) in a partial hospitalization program
  Interventions: Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in Children and Adolescents

INTERVENTIONS:
Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in Children and Adolescents — The Unified Protocols for Transdiagnostic Treatment of Emotional Disorders in Children and Adolescents (UP-C and UP-A) are transdiagnostic, behavioral interventions for youth with emotional disorders, including anxiety, depression, obsessive-compulsive disorders, and irritability.

SUMMARY:
The purpose of this study is to examine patient effectiveness outcomes of a transdiagnostic treatment for youth emotional disorders, implemented in a partial hospitalization program (PHP). Participants will be youth between ages 6 to 17 and their families, as well as clinicians, participating in the PHP program at Children's Hospital Colorado. Additionally, the research team will study modifications to the transdiagnostic intervention that are required to feasibly and effectively deliver it in a PHP setting.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patient participant involves:

* youth between the ages of 6 and 17
* participation in treatment in the Children's Hospital Colorado (CHCO) PHP program
* presence of at least one caregiver available and willing to participate in the study.

Inclusion criteria for clinician participants involves:

--psychologist, licensed master's-level clinician (i.e., "behavioral health clinician"), or unlicensed "behavioral health specialist" providing clinical services through the CHCO Partial Hospitalization Program during the period of study enrollment

Exclusion Criteria:

Patients will be excluded from the study if:

* they are a ward of the state
* are not enrolled in the Children's Hospital Colorado PHP program.

Clinicians will be excluded from the study if:

--they are not providing clinical services through the Children's Hospital Colorado PHP program

Ages: 6 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be youth and parents recruited from the partial hospitalization program at Children's Hospital Colorado.
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Client satisfaction with treatment, as measured by the Client Satisfaction Questionnaire-8 (CSQ-8) at post-treatment | 2 month
  The CSQ-8 is an 8-item, self and parent-report measure of satisfaction with treatment services. Total scores range from 8 to 32, with higher scores indicating greater satisfaction with treatment services.
Client satisfaction with treatment, as measured by the Client Satisfaction Questionnaire-8 (CSQ-8) at 1 Month follow up | 2 month
  The CSQ-8 is an 8-item, self and parent-report measure of satisfaction with treatment services. Total scores range from 8 to 32, with higher scores indicating greater satisfaction with treatment services.
Change in anxiety symptoms, as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric and Parent Proxy Anxiety Short Forms, Version 2.0 | Baseline, up to 2 month
  The PROMIS Pediatric and Parent Proxy Anxiety Short Form, Version 2.0 is an 8-item measuring assessing anxiety symptoms in youth. Total scores range from 8 to 40, with higher scores indicating greater anxiety symptoms.
Change in depression symptoms, as measured by the PROMIS Pediatric and Parent Proxy Depressive Symptoms Short Forms, Version 2.0 | Baseline, up to 2 month
  The PROMIS Pediatric and Parent Depressive Symptoms Short Form, Version 2.0 is a 6-item measuring assessing depressive symptoms in youth. Total scores range from 6 to 30, with higher scores indicating greater anxiety symptoms.
Change in emotional reactivity, as measured by the Emotion Dysregulation Inventory--Reactivity Short Form (EDI-R) | Baseline, up to 2 month
  The EDI-R is a 7-item, parent report measure of emotional reactivity in youth. Total scores range from 0 to 35, with higher scores indicating greater emotional reactivity.
Change in functional impairment, as measured by the Brief Impairment Scale (BIS) | Baseline, up to 2 month
  The BIS is a 23-item, parent report measure of functional impairment related to psychiatric symptoms in youth. Total scores range from 0 to 69, with higher scores indicating greater functional impairment.
Change in symptoms of disruptive and oppositional behavior, as measured by the Disruptive Behavior Rating Scale (DBRS) | Baseline, up to 2 month
  The DBRS is an 8-item, parent report measure assessing symptoms of disruptive behaviors/oppositional defiant disorder in youth. Total scores range from 0 to 24, with higher scores indicating more disruptive/oppositional behaviors.
Change in anxiety sensitivity, as measured by the Childhood Anxiety Sensitivity Index (CASI) | Baseline, up to 2 month
  The CASI is an 18-item self-report measure assessing fear of physiological symptoms of anxiety in youth. Total scores range from 18 to 56, with higher scores indicating greater anxiety sensitivity.
Change in distress intolerance, as measured by the Distress Intolerance Index for Youth (DIIY) | Baseline, up to 2 month
  The DIIY is a 10-item, self and parent-report measure assessing youth perceived inability to tolerate negative emotional states and experiential discomfort. Total scores range from 10 to 50, with higher scores indicating greater distress intolerance.

SECONDARY OUTCOMES:
Change in parental accommodation of youth emotional disorder symptoms, as measured by the Family Accommodation Scale (FAS-E), adapted for youth emotional disorders symptoms | Baseline, up to 2 month
  The FAS-E is a 9-item parent-report measure assessing family accommodation of emotions. Total scores range from 0 to 36, with higher scores indicating greater parent accommodation of emotion.
Change in positive and negative parenting behaviors, as measured by the Alabama Parenting Questionnaire--Short Form (APQ-S) | Baseline, up to 2 month
  The APQ-S is a 9-item, parent-report measure that yields three subscales ("Positive Parenting;" "Inconsistent Discipline," and "Poor Supervision"). Scores on each subscale range from 3 to 15. Higher scores on the Positive Parenting subscale indicate greater use of positive parenting strategies, higher scores on the Inconsistent Discipline scale indicate more inconsistent use of discipline techniques, and higher scores on the Poor Supervision scale indicate poorer parental supervision of youth.
Change in parents' perceived self-efficacy in parenting their child, as measured by the Parenting Sense of Competence--Parenting Self Efficacy Scale (PSOC) | Baseline, up to 2 month
  The PSOC is a 7-item measure assessing parents' perceived parenting self-efficacy. Total scores range from 7 to 42, with higher scores indicating greater parenting self-efficacy.
Change in youth cognitive reappraisal, as measured by the Emotion Regulation Questionnaire for Children and Adolescents--Reappraisal Scale (ERQ-CA) | Baseline, up to 2 month
  The ERQ-CA Reappraisal subscale is a 6-item measure assessing youth reappraisal, or the extent to which youth are able to change their thinking about situations that elicit emotions. Total scores range from 0 to 24, with higher scores indicating greater use of reappraisal.
Change in youth perceived self-efficacy, as measured by the PROMIS Self Efficacy scale | Baseline, up to 2 month
  The PROMIS Self Efficacy scale is a 10-item, self-report measure assessing general self-efficacy, or an individual's belief in their capacity to manage daily stressors and have control over meaningful events. Total scores range from 10 to 50, with higher scores indicating greater perceived self-efficacy.
Number of modifications made to the transdiagnostic treatment protocol, as measured by the Modification and Adaptation Checklist (MAC) | Up to 2 months
  The MAC is a 13-item checklist (including clinician self-report and observer report versions) intended to assist in tracking modifications made to an evidence-based treatment protocol. Adaptations and modifications will be tracked during 25% of treatment sessions. Total number of modifications will be summed.
Type of modifications made to the transdiagnostic treatment protocol, as measured by the Modification and Adaptation Checklist (MAC) | Up to 2 months
  The MAC is a 13-item checklist (including clinician self-report and observer report versions) intended to assist in tracking modifications made to an evidence-based treatment protocol. Adaptations and modifications will be tracked during 25% of treatment sessions. Types of modifications will be summarized categorically, and number of modifications of each type will be reported.
Fidelity to the transdiagnostic treatment protocol, as measured by the UP-C Adherence and Competency Checklist, Observer and Clinician Self-Report version | Up to 2 months
  The UP-C Adherence and Competency Checklist is a tool designed to facilitate tracking of the delivery of core treatment components during therapy sessions. 25% of group therapy sessions will be coded by an observer and by clinicians delivering the intervention, and proportion of core elements delivered will be calculator. Inter-rater reliability among reporters will also be calculated. Score range: 0-170 (scored on a three-point scale) Higher scores indicate greater therapist competence and adherence to the treatment protocol. Scores are represented as percent adherence rather than total (e.g., 90% adherent).
Fidelity to the transdiagnostic treatment protocol, as measured by the UP-A Adherence and Competency Checklist, Observer and Clinician Self-Report version | Up to 2 months
  The UP-A Adherence and Competency Checklist is a tool designed to facilitate tracking of the delivery of core treatment components during therapy sessions. 25% of group therapy sessions will be coded by an observer and by clinicians delivering the intervention, and proportion of core elements delivered will be calculator. Inter-rater reliability among reporters will also be calculated. Score range: 0-170 (scored on a three-point scale). Higher scores indicate greater therapist competence and adherence to the treatment protocol. Scores are represented as percent adherence rather than total (e.g., 90% adherent).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah M Kennedy, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results reported in any published studies will be shared upon publication, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available immediately following publication and ending 5 years after publication.
Access Criteria: Researchers who provide a methodologically sound proposal or reason for accessing the data will be granted access.